CLINICAL TRIAL: NCT01823029
Title: Oxidative Stress and Inflammation Caused by Intravenous Iron in Crohn's Disease Patients With Iron Deficiency Anemia
Acronym: CD-AT1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Collaborators: Ministry of Health, China (Other Government)
Responsible Party: Principal Investigator, Zhu Weiming, vice director of General surgery institute, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CD-AT1
Record Dates: First submitted 2013-03-25; First posted 2013-04-04 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; intravenous iron; iron deficiency anaemia; Oxidative Stress; inflammation
MeSH Terms: conditions — Crohn Disease; Anemia, Iron-Deficiency; Inflammation | interventions — Erythropoietin; Enteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- erythropoietin,injection of iron and enteral nutrition (Experimental): The patients receive treatment of erythropoietin,injection of iron and enteral nutrition.
  Interventions: Drug: erythropoietin; Drug: enteral nutrition.; Drug: injection of iron
- erythropoietin and enteral nutrition. (Experimental): The patients receive treatment of erythropoietin and enteral nutrition.
  Interventions: Drug: erythropoietin; Drug: enteral nutrition.

INTERVENTIONS:
Drug: erythropoietin
Drug: enteral nutrition.
Drug: injection of iron
  Arms: erythropoietin,injection of iron and enteral nutrition

SUMMARY:
Extra iron may not be necessary in the treatment of iron deficiency anemia in Crohn's Disease;Oxidative Stress and Inflammation may be Caused by Intravenous Iron in Crohn's Disease Patients With Iron Deficiency Anemia.

DETAILED DESCRIPTION:
Anemia is one of the commonest extra-intestinal manifestations of Crohn's disease (CD) with a prevalence ranging from 6.2% up to 73.7%.Compared with other complications,it has been subestimated and received less attention from gastroenterologists, although,which is frequently associated with a reduced quality of life.What's more,there were not appropriate strategies for the adequate treatment of anaemia in CD either.

The anaemia in CD is caused by several factors, such as iron, folic acid or B12 deficiency, treatment with immunosuppressive drugs or sulfasalazine-induced hemolysis, and anemia of chronic disease, of which iron deficiency was one of the most important mechanisms. Additionally, erythropoietin(EPO) levels in chronic disease anemia are generally higher than in normal subjects.However, in CD anemic patients this EPO increase is inadequate in relation to the degree of anemia.Thus, in the treatment of iron deficiency anemia (IDA) in CD,EPO and iron supplementation are very common.Because intravenous(IV) iron is more effective and better tolerated than oral iron and is to be considered in patients with severe anemia (Hb<10.0 g/dL), with intolerance or inadequate response to oral iron and/or those with active IBD. Intravenous iron administration is the route of choice when simultaneous treatment with erythropoiesis stimulat-ing agents (ESA) is considered.

But parenteral iron formulations have potential toxic effects such as triggering oxidative reactions and inflammatory reactions that may be very disadvantageous to CD patients. Free iron may provoke formation of free oxygen radicals. Although complex carbohydrate structures that cover free iron may alleviate this oxidative and inflammatory potential,it cannot be completely blocked. These suggest that parenteral iron could be a "double-edged sword" with the hematologic beneﬁts (increase in hemoglobin [Hb]) on the one hand, and with the risk of enhancement of systemic inﬂammation and oxidative stress on the other.

Although the oxidative potential of intravenous iron (IVI) has been studied extensively,there have been no studies about the effects of parenteral iron therapy on oxidative stress and inflammatory markers in the CD population. In this study, we compared different types and schedules of iron compounds for their effects on serum inflammatory-oxidative stress indices.

ELIGIBILITY:
Inclusion Criteria:

* Subjects should have a definitive diagnosis of Crohn's disease, based on WHO criteria
* Males and females ≥ 18 years old, including women who are not pregnant or lactating at the time of enrollment.
* Subjects should have a CDAI score <150 at week 0
* Able to swallow tablets
* Are capable of providing written informed consent and obtained at the time of enrollment
* Willing to adhere to the study visit schedule and other protocol requirements.
* Subjects should have the hemoglobin： male patients<130g/L，female patients<120g/L.

Exclusion Criteria:

* Bacterial,viral or other microbial infection(including HIV)
* Needing orally administered corticosteroids for the treatment of other diseases. Inhaled or dermatologic preparations are acceptable.
* Previous or current use of infliximab.
* current use of prescription doses or chronic/frequent use of NSAIDs
* Treatment with narcotic pain medications. (Anti-diarrheal agents such as loperamide and diphenoxylate are permitted)
* History of pancreatitis, except for subjects with a known but removed cause(such as gallstone pancreatitis)
* History of abnormal liver function tests, including AST or ALT >1.5 times upper limit of normal, alkaline phosphatase >2 times upper limit of normal, total bilirubin >2.5 mg/dL at screening (or within the previous 6 months, if known)
* History of malignancy
* Women who are pregnant or lactating at the time of enrollment, or who intend to be during the study period.
* Participation in other clinical trial within the past 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 387 (Actual)
Dates: Start 2012-11; Primary Completion 2013-07 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
haemoglobin raise to norm or not. | at 0 week, the first week, the second week, the third week, the fourth week

SECONDARY OUTCOMES:
The change of haematological inflammation marker(CRP,ESR,IL-10,IL-6,TNF-ａ,IL-1β) | at 0 week, the first week, the second week, the third week, the fourth week
The change of haematological oxidative stress indicators(SOD,GSH-px and MDA) | at 0 week, the first week, the second week, the third week, the fourth week
The change of patients'IBDQ and CDAI. | at 0 week and the fourth week
relapse of anaemia | 12 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: wei ming zhu, PhD,MD, Principal Investigator — General Surgery Institute,Jinling Hospital,Nanjing,Jiangsu,China
Locations (1):
- General Surgery Institute,Jinling Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Kulnigg S, Gasche C. Systematic review: managing anaemia in Crohn's disease. Aliment Pharmacol Ther. 2006 Dec;24(11-12):1507-23. doi: 10.1111/j.1365-2036.2006.03146.x. PMID 17206940
- [Background] Bergamaschi G, Di Sabatino A, Albertini R, Ardizzone S, Biancheri P, Bonetti E, Cassinotti A, Cazzola P, Markopoulos K, Massari A, Rosti V, Porro GB, Corazza GR. Prevalence and pathogenesis of anemia in inflammatory bowel disease. Influence of anti-tumor necrosis factor-alpha treatment. Haematologica. 2010 Feb;95(2):199-205. doi: 10.3324/haematol.2009.009985. Epub 2009 Oct 8. PMID 19815838
- [Background] Goodhand JR, Kamperidis N, Rao A, Laskaratos F, McDermott A, Wahed M, Naik S, Croft NM, Lindsay JO, Sanderson IR, Rampton DS. Prevalence and management of anemia in children, adolescents, and adults with inflammatory bowel disease. Inflamm Bowel Dis. 2012 Mar;18(3):513-9. doi: 10.1002/ibd.21740. Epub 2011 May 20. PMID 21604328
- [Background] Reinisch W, Staun M, Bhandari S, Munoz M. State of the iron: how to diagnose and efficiently treat iron deficiency anemia in inflammatory bowel disease. J Crohns Colitis. 2013 Jul;7(6):429-40. doi: 10.1016/j.crohns.2012.07.031. Epub 2012 Aug 20. PMID 22917870
- [Background] Ott C, Liebold A, Takses A, Strauch UG, Obermeier F. High prevalence but insufficient treatment of iron-deficiency anemia in patients with inflammatory bowel disease: results of a population-based cohort. Gastroenterol Res Pract. 2012;2012:595970. doi: 10.1155/2012/595970. Epub 2012 Jul 30. PMID 22899905
- [Background] Noskova KK, Lishchinskaia AA, Parfenov AI, Kniazev OV, Varvanina GG, Drozdov VN. [Risk of development of clinical and pathogenetic features of anemia on the background of basic therapy of inflammatory bowel disease]. Eksp Klin Gastroenterol. 2011;(10):12-7. Russian. PMID 22629693
- [Background] Voegtlin M, Vavricka SR, Schoepfer AM, Straumann A, Voegtlin J, Rogler G, Ballabeni P, Pittet V, Buser A, Fried M, Beglinger C; Swiss IBD Cohort Study. Prevalence of anaemia in inflammatory bowel disease in Switzerland: a cross-sectional study in patients from private practices and university hospitals. J Crohns Colitis. 2010 Dec;4(6):642-8. doi: 10.1016/j.crohns.2010.07.008. Epub 2010 Aug 12. PMID 21122574
- [Background] Katsanos KH, Tatsioni A, Natsi D, Sigounas D, Christodoulou DK, Tsianos EV. Recombinant human erythropoietin in patients with inflammatory bowel disease and refractory anemia: a 15-year single center experience. J Crohns Colitis. 2012 Feb;6(1):56-61. doi: 10.1016/j.crohns.2011.07.004. Epub 2011 Aug 17. PMID 22261528
- [Background] Jian J, Yang Q, Dai J, Eckard J, Axelrod D, Smith J, Huang X. Effects of iron deficiency and iron overload on angiogenesis and oxidative stress-a potential dual role for iron in breast cancer. Free Radic Biol Med. 2011 Apr 1;50(7):841-7. doi: 10.1016/j.freeradbiomed.2010.12.028. Epub 2010 Dec 28. PMID 21193031
- [Background] Fishbane S, Kowalski EA. The comparative safety of intravenous iron dextran, iron saccharate, and sodium ferric gluconate. Semin Dial. 2000 Nov-Dec;13(6):381-4. doi: 10.1046/j.1525-139x.2000.00104.x. PMID 11130261